CLINICAL TRIAL: NCT02048956
Title: 8-weeks Hydrotherapy Intervention in Patients With Knee Osteoarthritis.
Brief Title: Hydrotherapy Intervention in Elderly With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DF0049UG
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; hydrotherapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrotherapy intervention (Experimental): 30 people will be recruited in order to the inclusion criteria for the study and they will receive an hydrotherapy intervention.
  Interventions: Other: Hydrotherapy intervention
- Control group (Active Comparator): 30 people will be recruited and included in this control group. The are not going to receive hydrotherapy treatment, only the treatment they receive as usual.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Hydrotherapy intervention — Participants randomized to the exercise programme received a training in a swimming pool focused on dance therapy.
  Other Names: Exercise program; Swimming pool training
  Arms: Hydrotherapy intervention
Other: Control group — Standard exercises of hydrotherapy
  Other Names: Standard hydrotherapy intervention
  Arms: Control group

SUMMARY:
Knee osteoarthritis is a common condition characterized by pain and functional disability in older people. Prevalence increases with age and is more frequent in older women. The aim of this study was to assess the effects of an 8-weeks hydrotherapy training with elastic bands on pain and functional disability in old people with knee osteoarthritis.

DETAILED DESCRIPTION:
The main symptoms of knee osteoarthritis are pain and functional disability. These symptoms are caused by a progressive loss and deterioration of articular cartilage with reactive new bone formation at the joint's surface and margins involving articular cartilage, soft tissues and bone damage. Many treatment programs have been developed, including medication with nonsteroidal anti-inflammatory drugs, physical modalities, and therapeutic exercises. It is hypothesized that a hydrotherapy treatment during 8 weeks would benefit patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* confirmed clinical diagnosis of knee osteoarthritis

Exclusion Criteria:

* total knee arthroplasty
* inability to co-operate or follow instructions.
* a major neurological disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in pain pressure threshold | baseline, 8 weeks
  The pain pressure threshold is defined as the minimum amount of pressure necessary to induce pain or tenderness . It was measured using a pressure algometer (Somedic AB, Sweden), which is a device with a 1 cm diameter rubber disc at the end on quadriceps muscle.

SECONDARY OUTCOMES:
Changes in lower extremity strength | baseline, 8 weeks
  Changes in the strength of lower limbs is going to be assessed using the Stairs Climbing Test. This test assesses the ability to ascend and descend a flight of stairs, as well as lower extremity strength, power, and balance.
Dual task | baseline, 8 weeks
  Dual task is going to be measured using the Timed Up & Go. It assesses basic mobility skill as well as strength, balance, and agility.
Functional ability | baseline, 8 weeks
  Functional ability was assessed by the Western Ontario and McMaster Universities Osteoarthritis Index. Higher scores on the this questionnaire represent greater limitations in function.
Changes in balance | baseline, 8 weeks
  The in balance after the treatment is going to be assessed using the single leg stance. This is a clinical tool that is often used to assess balance and postural steadiness. Subjects are asked to lift one leg off the floor based on their preference and keep the leg raised as long as possible without touching the other leg or the floor

OTHER OUTCOMES:
Quality of sleep | baseline, 8 weeks
  Quality of sleep was assessed by Pittsburgh Sleep Quality Index, a self-reported questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of health Sciences. University of Granada, Granada, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided